CLINICAL TRIAL: NCT03031522
Title: Molecular Imaging to Identify EGFR-TKIs Benefit Non-small Cell Lung Carcinoma Patients
Brief Title: EGFR Molecular Classification In Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yingying Sun, Chief, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14006
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-01

CONDITIONS: Molecular Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 18F-IRS : EGFR+ Patients (Experimental): Patients in this group had EGFR-activating mutant tumors and did not receive any treatment before this study.
  Interventions: Radiation: 18F-IRS
- 18F-IRS :post-TKI EGFR+ Patients (Experimental): Patients with EGFR-activating mutant tumors were receiving EGFR-TKIs during this study .
  Interventions: Radiation: 18F-IRS
- 18F-IRS:post-chemo EGFR+ (Experimental): 18F-IRS:post-chemo EGFR+ Patients with EGFR-activating mutant tumors were receiving chemotherapy during this study.
  Interventions: Radiation: 18F-IRS
- 18F-IRS:EGFR wild type (Experimental): Patients in this group had EGFR wild-type tumors and did not receive any treatment before this study.
  Interventions: Radiation: 18F-IRS
- 18F-IRS:post-chemo EGFR wild type (Experimental): Patients in this group had EGFR wild-type tumors and were receiving chemotherapy during this study.
  Interventions: Radiation: 18F-IRS
- 18F-IRS:unknown EGFR mutational status (Experimental): Patients without the EGFR mutational status measurement results and did not receive any treatments were classified in this group
  Interventions: Radiation: 18F-IRS

INTERVENTIONS:
Radiation: 18F-IRS — According to experiment, 18F-IRS was non-toxic and stable in serum.

SUMMARY:
The investigators developed 18F-IRS as a targeted molecular imaging agent for noninvasive and repeatable detecting EGFR-activating mutational status.

DETAILED DESCRIPTION:
The goal of investigators were to evaluate the use of 18F-IRS as a novel PET/CT radiotracer to monitor EGFR-activating mutational status and identify EGFR-TKIs benefit NSCLC patients. the investigators want to evaluated the use of 18F-IRS in lung cancer imaging in adult NSCLC patients with different EGFR mutational status of primary and metastatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* 18 years or older
* A life expectancy of at least 12 weeks
* Presence of a malignant lesion within the chest of at least 0.5 cm diameter as measured by computed tomography (CT)
* Written informed consent

Exclusion Criteria:

* Claustrophobia
* Pregnancy
* Metal implants in the thorax

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
tumor SUVmax value of 18F-IRS PET/CT Imaging | at time of imaging
  To quantify the accumulation, a volume of interest using a 3-D sphere, was placed over the primary lung tumor, lymph nodes and distant metastases avoiding necrosis, blood vessels and normal lung tissue as much as possible on a workstation (Advantage Workstation 4.6; GE Healthcare). The maximum standard uptake value (SUVmax) normalized to body weight (kBq/mL) was calculated within the region of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Baozhong Shen, M.D., Study Chair — The Fourth Hospital of Harbin Medical University
Locations (1):
- TOF-PET/CT/MR center of the Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided